CLINICAL TRIAL: NCT05118607
Title: The Use of Microcurrent and Low Current Bioelectrical Stimulation in the Treatment of Post-prostatectomy Erectile Dysfunction
Brief Title: The Use of Bioelectrical Stimulation in the Treatment of Post-prostatectomy Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Cristiane Carboni, Professor, Federal University of Health Science of Porto Alegre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02718918.1.0000.5221
Record Dates: First submitted 2021-11-02; First posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Erectile Dysfunction Following Radical Prostatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (IG1) (Other): application of low intensity transcutaneous penile electrical stimulation for 45 minutes using frequency
  Interventions: Device: IG1

INTERVENTIONS:
Device: IG1 — application of low intensity transcutaneous penile electrical stimulation for 45 minutes using frequency.

SUMMARY:
Erectile dysfunction (ED) affects up to 20% of men and is a growing problem with advancing age. There are many causes that contribute to ED, including the concomitant use of prescription drugs for health problems, including hypertension, or diseases such as diabetes. causes an up-regulation or increased local tissue expression of these proteins. This study follows the demonstration of the effectiveness of using BES in the treatment of ED. The aim of this study will be to examine the potentially additive effect of adding a third arm to the previous protocol to include the addition of 4 new target proteins to VEGF, including endothelial nitric oxide (eNOS), stromal-derived factor 1 (SDF-1), insulin-like growth factor (IGF) and follistatin.

DETAILED DESCRIPTION:
For this randomized clinical trial, 10 patients from a private Urology clinic will be selected. Each patient will serve as their own two-month documentation control using the validated IIEF-5 and EHS questionnaires. The intervention period will last 8 weeks. And 6 months of follow-up after the end of treatment to see how long the benefit lasts without continued treatment. The assessment will be carried out before the intervention period (pre-intervention) and after the intervention period (post-intervention and follow-up) for all participants. All patients who, after medical consultation, are diagnosed with erectile dysfunction and who meet the inclusion criteria will be included in the study.

Erectile function will be assessed using the validated questionnaire IIEF-5. The instrument will be completed by a blind researcher and the technique will be applied by a physiotherapist trained in the area.

Erectile dysfunction (ED) was defined as the inability to achieve and/or maintain sufficient penile erection for satisfactory sexual performance 11 for at least 6 months, accompanied by an IIEF5 questionnaire score of less than 22 points.

The patients were in the supine position, in a lithotomy position. They will undergo trichotomy at the site of placement of the self-adhesive surface electrodes. Each patient will have their own pair of electrodes that will be used until the end of therapy, and they will be discarded after the end of the sessions. The intervention will consist of the application of low intensity transcutaneous penile electrical stimulation for 45 minutes using frequency.

ELIGIBILITY:
Inclusion Criteria:

Male patient, aged 40 to 75 years, with a stable marital relationship (6 months) Diagnosis of post-prostatectomy erectile dysfunction (IIEF5 score less than 22)

Exclusion Criteria:

Neurogenic ED (spinal injury, Parkinson, MS) Hypogonadism (total testosterone < 300 ng/dl) Decompensated diabetes mellitus (Fasting Glucose>200 and/or Glycated Hemoglobin>8%) Decompensated systemic arterial hypertension (SBP > 160 and/or DBP >100 Morbid obesity Use of vacuum device smokers Diagnosis of coronary artery disease and/or cerebrovascular disease Impossibility of understanding the objectives, study technique and informed consent cognitive deficit

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — erectile dysfunction
Enrollment: 10 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
The present study aims to evaluate the effect of BES on post-prostatectomy ED using the International Index of Erectile Function-5 (IIEF-5) questionnaire and the Erection hardness Score (EHS) questionnaire. | 1 year
  The present study aims to evaluate the effect of BES on post-prostatectomy ED using the International Index of Erectile Function-5 (IIEF-5) questionnaire and the Erection hardness Score (EHS) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane Carboni, Principal Investigator — Professor
Locations (1):
- Mundo do Assoalho Pélvico, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided